CLINICAL TRIAL: NCT02694471
Title: CB147 - Physical Activity and Nutrition for Quality Ageing
Brief Title: Effect of 14 Day Bed Rest on Health Outcomes in Young and Older Participants
Acronym: BEDREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: University of Trieste (Other); University of Udine (Other); University of Padova (Other); Università degli Studi di Ferrara (Other); University of Nottingham (Other); DLR German Aerospace Center (Other); Izola General Hospital (Other); National Institute of Public Health, Slovenia (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PANGEA
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Muscular Atrophy
Keywords: Ageing; Physical inactivity; Functional decline; Reconditioning
MeSH Terms: conditions — Muscular Atrophy; Sedentary Behavior | interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Old group (Experimental): 16 old participants (55-65 years) were included in physical inactivity or bed rest with supervised recovery intervent and underwent 14-day of bed rest. Bed rest was followed by 28-day recovery. During the bed rest participants will remain 24-hour horizontal with all daily activities performed lying in a bed. No social isolation will be forced. During the recovery participants will 3-times weekly per 75 minutes perform guided exercises to achieve baseline level.
  Interventions: Behavioral: physical inactivity or bed rest with supervised recovery
- Young group (Active Comparator): 7 young participants (18-30 years) were included in physical inactivity or bed rest with supervised recovery intervent and underwent 14-day of bed rest. Bed rest was followed by 28-day recovery. During the bed rest participants will remain 24-hour horizontal with all daily activities performed lying in a bed. No social isolation will be forced. During the recovery participants will 3-times weekly per 75 minutes perform guided exercises to achieve baseline level.
  Interventions: Behavioral: physical inactivity or bed rest with supervised recovery

INTERVENTIONS:
Behavioral: physical inactivity or bed rest with supervised recovery — All (older and younger) participants underwent 14 day of horizontal bed rest with all 24 hour daily activities were performed lying in a bed. Maximal one pillow was allowed. 28-day supervised recovery was performed 3 times weekly for 75 minutes/session.

SUMMARY:
This investigation aimed to compare the response of older adult and young men to 14 day bed-rest and subsequent 28 day rehabilitation. Sixteen older (OM: 55-65 years) and seven young men (YM: 18-30 years) were exposed to 14-day bed rest (BR) followed by 14-day rehabilitation (R), and 400-day of R. Quadriceps muscle volume, force and explosive power of leg extensors, single fiber isometric force, peak aerobic power, gait stride length, and several metabolic were measured before and after BR and after R.

DETAILED DESCRIPTION:
Twenty-three healthy men, of which 7 young (YM; aged 18-30 years) and 16 older adults (OM; aged 55-65 years) were recruited for the study. All participants underwent medical examination and routine blood and urine analysis. Exclusion criteria were: smoking; regular alcohol consumption; ferromagnetic implants; history of deep vein thrombosis with D-dimer > 500 μg·L-1; acute or chronic skeletal, neuromuscular, metabolic and cardiovascular disease conditions; pulmonary embolism. Participants were informed of the purpose, procedures and potential risk of the study before signing the informed consent. The study was performed in accordance with the ethical standards of the 1964 Declaration of Helsinki and was approved by the National Ethical Committee of the Slovenian Ministry of Health on April 17, 2012.

The study was conducted in controlled medical environment of the Orthopedic Hospital of Valdoltra, Slovenia. The participants were housed in standard air conditioned hospital rooms and were under constant surveillance with 24-hour medical care. For 14 days, the participants performed all daily activities in bed and received eucaloric controlled meals three times a day. Dietary energy requirements were designed for each subject multiplying resting energy expenditure by factors 1.2 and 1.4 in BR and ambulatory period, respectively. The resting energy expenditure was calculated as done in previous studies. The macronutrient food content set at 60% of carbohydrates, 25% fat, and 15% of proteins, according to the scheme of the so called "mediterranean diet" and adopted also in previous bed rest protocols. Energy balance was checked weekly by fat mass assessment. The daily protein intake was 1.1-1.25 g kg-1 in both groups, in BR and recovery period respectively, except the subgroups of OM who received a supplementation (see below).

After the BR, participants underwent a rehabilitation protocol (R) that consisted of 4-week supervised multimodal exercise program with 3 sessions per week. In each session, participants performed 12-minute warm-up, 15-20 minutes of balance and strength training, and 20-30 minutes of endurance training.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 28 kg/m2
* Short physical performance battery score >= 9

Exclusion Criteria:

* smoking;
* regular alcohol consumption;
* ferromagnetic implants;
* history of deep vein thrombosis with D-dimer > 500 μg·L-1;
* acute or chronic skeletal, neuromuscular, metabolic and cardiovascular disease conditions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps muscle volume (young vs. old) after 14-day bed rest | At baseline and after 14-day bed rest and on 14th day of recovery
  Using MRI continous screening of single leg was performed
Change in diameter of single fibre contractions (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  Biopsy samples were obtained from vastus lateralis muscles
Change in peak aerobic power (VO2max) (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  graded cycling on sitting ergometer until exhaustion

SECONDARY OUTCOMES:
Change in peak knee extensor force (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  Estimated from single leg isometric maximal voluntary contraction
Change in lower limb explosive power (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  estimated from bilateral efforts on explosive ergometer (EXER)
Change in gait stride length (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th and 400th day of recovery
  Walking through the food placement detection system
Change in insulin sensitivity (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  collected hourly for 6 hours after standard meal load as a measure of insulin sensitivity index
Change in area-under-the curve (AUC) of triglycerides plasma concentration (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  collected hourly for 3 hours after standard meal load
Change in N-telopeptide (young vs. old) after 14-day bed rest | baseline, during and after 14-day bed rest and during first 14 day of recovery
  From urine collection
Change in C-telopeptide (young vs. old) after 14-day bed rest | baseline, during and after 14-day bed rest and during first 14 day of recovery
  From urine collection
Change is contraction time (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  From Tensiomyographic response in vastus lateralis
Change in force of single muscle fibre contraction (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  Biopsy samples were obtained from vastus lateralis muscles
Change in specific force of single muscle fibre contraction (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  Biopsy samples were obtained from vastus lateralis muscles
Change in velocity of single muscle fibre contraction (young vs. old) after 14-day bed rest | baseline and after 14-day bed rest and on 14th day of recovery
  Biopsy samples were obtained from vastus lateralis muscles

CONTACTS AND LOCATIONS:
Overall Officials: Rado Pišot, PhD, Principal Investigator — University of Primorska, Slovenia
Locations (1):
- Orthopaedic Hospital Valdoltra, Ankaran, Slovenia

IPD SHARING:
Plan to Share IPD: No
The data is shared among partners for various publications

REFERENCES:
- [Result] Pisot R, Marusic U, Biolo G, Mazzucco S, Lazzer S, Grassi B, Reggiani C, Toniolo L, di Prampero PE, Passaro A, Narici M, Mohammed S, Rittweger J, Gasparini M, Gabrijelcic Blenkus M, Simunic B. Greater loss in muscle mass and function but smaller metabolic alterations in older compared with younger men following 2 wk of bed rest and recovery. J Appl Physiol (1985). 2016 Apr 15;120(8):922-9. doi: 10.1152/japplphysiol.00858.2015. Epub 2016 Jan 28. PMID 26823343
- [Result] Jurdana M, Jenko-Praznikar Z, Mohorko N, Petelin A, Jakus T, Simunic B, Pisot R. Impact of 14-day bed rest on serum adipokines and low-grade inflammation in younger and older adults. Age (Dordr). 2015 Dec;37(6):116. doi: 10.1007/s11357-015-9848-z. Epub 2015 Nov 13. PMID 26564239
- [Result] Marusic U, Kavcic V, Giordani B, Gerzevic M, Meeusen R, Pisot R. Computerized spatial navigation training during 14 days of bed rest in healthy older adult men: Effect on gait performance. Psychol Aging. 2015 Jun;30(2):334-340. doi: 10.1037/pag0000021. Epub 2015 May 4. PMID 25938245
- [Result] Goswami N, Kavcic V, Marusic U, Simunic B, Rossler A, Hinghofer-Szalkay H, Pisot R. Effect of computerized cognitive training with virtual spatial navigation task during bed rest immobilization and recovery on vascular function: a pilot study. Clin Interv Aging. 2015 Feb 10;10:453-9. doi: 10.2147/CIA.S76028. eCollection 2015. PMID 25709419